CLINICAL TRIAL: NCT03437330
Title: Empagliflozin Effect on Glucose Toxicity in Type 2 Diabetes Patients - a Randomized, Open-label, Controlled, Parallel Group, Exploratory Study
Brief Title: Empagliflozin Effect on Glucose Toxicity
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oxidise
Record Dates: First submitted 2017-12-21; First posted 2018-02-19 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — empagliflozin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Jardiance®) (Experimental): Dose/frequency: 10 mg once daily for 12 weeks Route of administration: oral
  Interventions: Drug: Empagliflozin (Jardiance®)
- Insulin Glargine (Lantus®) (Active Comparator): Thus, insulin glargine doses should be adapted as follows:
  FBG 6-7 mmol/L: +2 IU FBG 7-8 mmol/L: +3 IU FBG > 8 mmol/L: +5 IU
  Interventions: Drug: Insulin Glargine (Lantus®)

INTERVENTIONS:
Drug: Empagliflozin (Jardiance®) — Empagliflozin Dose/frequency: 10 mg once daily for 12 weeks Route of administration: oral Reference group: Insulin glargine (Lantus®) Dose/frequency: see below FBG 6-7 mmol/L: +2 IU (stop when FBG is reduced by 0.5 mmol/L or documented hypoglycemia < 3.9 mmol/L occurs) FBG 7-8 mmol/L: +4 IU (stop when FBG is reduced by 1.0 mmol/L or documented hypoglycemia < 3.9 mmol/L occurs) FBG > 8 mmol/L: +6 IU (stop when FBG is reduced by 1.5 mmol/L or documented hypoglycemia < 3.9 mmol/L occurs)
  Arms: Empagliflozin (Jardiance®)
Drug: Insulin Glargine (Lantus®) — insulin glargine shall be titrated according to the following scheme: If FBG 6-7 mmol/L: reduce fasting glucose by 0.5 mmol/L If FBG 7-8 mmol/L: reduce fasting glucose by 0.75 mmol/L
  If FBG 8-9 mmol/L: reduce fasting glucose by 1.0 mmol/L Thus, insulin glargine doses should be adapted as follows:
  FBG 6-7 mmol/L: +2 IU (stop when FBG is reduced by 0.5 mmol/L or documented hypoglycemia < 3.9 mmol/L occurs) FBG 7-8 mmol/L: +3IU (stop when FBG is reduced by 0.75 mmol/L or documented hypoglycemia < 3.9 mmol/L occurs) FBG > 8 mmol/L: +5 IU (stop when FBG is reduced by 1.0mmol/L or documented hypoglycemia < 3.9 mmol/L occurs)
  Arms: Insulin Glargine (Lantus®)

SUMMARY:
Empagliflozin effect on glucose toxicity in type 2 diabetes patients - a randomized, open-label, controlled, parallel group, exploratory study

DETAILED DESCRIPTION:
The EMPA-REG outcome trial showed that empagliflozin on top of standard therapy for Type 2 diabetes mellitus (T2DM) resulted in superiority in terms of the primary composite cardiovascular endpoint (hazard ratio (1) = 0.86; 95% confidence interval [CI] 0.74-0.99; P value = 0.04), hospitalization for heart failure (-35%), cardiovascular mortality (-38%) and all-cause mortality (-32%, each p < 0.001) (2). This reduction in mortality is not fully explained by the reduction in HbA1c, body weight, waist circumference and blood pressure in the empagliflozin groups versus the placebo group. Differences in mode of action of empagliflozin compared to standard therapy might, thus, help to explain why empagliflozin was so efficient in reducing cardiovascular death.

The aim of the present study is to provide evidence for a reduction of skeletal muscle H2O2 levels, and consequently improvement in mitochondrial function, and restored methylation pattern of key transcription factors in skeletal muscle from patients with T2DM when treated with empagliflozin versus insulin glargine as the prototypical medication favoring glucose uptake into tissues. It is hypothesized that empagliflozin compared to insulin specifically reduces H2O2 concentrations in skeletal muscle of patients with T2DM, because it leads to excretion of glucose and lower glucose uptake in skeletal muscle (22), while insulin shifts the major part of excess glucose into skeletal muscle cells.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria before inclusion in the study:

* The informed consent form must be signed before any study specific tests or procedures are done
* Male or female patients aged between 40 and 70 years (including) at the first screening visit
* Patients diagnosed with T2DM
* HbA1c between 7-9% (including)
* Stable treatment with antidiabetic drugs over the last 4 weeks
* Accepted background medication:

  * Metformin up to 2000 mg per day and/or
  * DPP-IV inhibitors:

Linagliptin up to 5 mg per day Sitagliptin up to 100 mg per day Vildagliptin up to 100 mg per day Saxagliptin up to 5 mg per day

* Body mass index (BMI) between 25 and 40 kg/m2 (including)
* Ability to understand and follow study-related instructions
* No clinical relevant abnormalities during ECG and cardiac examinations

Exclusion Criteria:

Subjects are to be excluded from the study if they display any of the following criteria:

* Unstable Angina pectoris, myocardial infarction or stroke within 1 year before inclusion in the study
* History of atrial fibrillation
* Uncontrolled arterial hypertension (> 160/100 mmHg in three subsequent measurements - mean value)
* eGFR < 60 ml/min/1.73 m2
* Macroalbuminuria defined as ≥ 300 mg albumin / 24h urine
* Triglyceride > 250 mg/dl
* Genetic muscle disease
* Known coagulation disorder
* Treatment with anti-platelet therapy and anticoagulation which cannot be paused for medical reasons
* Treatment with anticoagulants within 7 days prior to the muscle biopsy
* Contraindications according to the local SmPC of Lantus® or Jardiance® (see Appendix 1)
* History of hypersensitivity to any of the study drugs or their ingredients or to drugs with similar structure or to the local anesthetic scandicaine or lidocaine
* Addiction or other diseases that preclude the patient from appropriately assessing the nature and scope as well as possible consequences of the clinical study
* Pregnant or breast-feeding women
* Women of childbearing potential unless women who meet the following criteria:

  * Post-menopausal (12 months natural amenorrhea or 6 months amenorrhea with serum follicle-stimulating hormone [FSH] > 40 U/mL)
  * Postoperatively (six weeks after bilateral ovariectomy with or without hysterectomy)
  * Regular and correct use of a contraceptive method with error rate <1% per year such as implants, depot injections, oral contraceptives or intrauterine devices
  * Sexual abstinence
  * Vasectomy of the partner
* Males must agree not to father a child and to refrain from donating semen or sperm while participating in the study and for 90 days following discontinuation from this study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Change in skeletal muscle H202 concentration between baseline and end of treatment (EoT) | 12 weeks
  The primary objective is to investigate the change in H2O2 concentration as a read out of reactive oxygen species (ROS) production in skeletal muscle biopsies from T2DM patients before and after treatment with empagliflozin or insulin glargine.

SECONDARY OUTCOMES:
Secondary objectives of the study are to evaluate the effect of empagliflozin and insulin glargine on glucose toxicity in skeletal muscle by investigating | 12 weeks
  Change in skeletal muscle mitochondrial function (O2consumption) between baseline and EoT
Change in skeletal muscle lipid peroxidation | 12 weeks
  Change in skeletal muscle lipid peroxidation between baseline and EoT
Change in 24-hour urinary excretion rate of 8-iso PGF2a | 12 weeks
  Change in 24-hour urinary excretion rate of 8-iso PGF2a between baseline and EoT
• Difference in DNA methylation pattern | 12 weeks
  • Difference in DNA methylation pattern between the treatment groups at EoT
Change in plasma FFA levels | 12 weeks
  Change in plasma FFA levels between baseline and end of trial

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital, Tübingen, Baden-Wurttemberg
  - German Diabetes Center, Leibniz-Center for Diabetes Research at the Heinrich-Heine-University Duesseldorf, Düsseldorf, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No